CLINICAL TRIAL: NCT03007953
Title: Palliative Care Interventions for Outpatients Newly Diagnosed With Lung Cancer: Phase II
Acronym: PCI2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRI 15-456
Record Dates: First submitted 2016-12-19; First posted 2017-01-02 (Estimated); Results first posted 2021-10-07 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Lung Cancer
Keywords: Palliative Care; Supportive Care
MeSH Terms: conditions — Lung Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): This is a nurse-led telephone-based program integrating palliative care into usual oncologic care for patients diagnosed within 2 months of any type and stage of lung cancer, who will receive therapy other than solely surgical resection. The intervention lasts for the duration of patients' primary lung cancer treatment (usually 3-4 months).
  Interventions: Behavioral: Palliative Care
- Usual Care (No Intervention): Subjects randomized to the usual care arm will receive medical oncology, radiation oncology, pulmonary, CT surgery, as indicated by the type and stage of cancer. At the completion of their primary lung cancer treatment, they will be disenrolled from the study.

INTERVENTIONS:
Behavioral: Palliative Care — Care delivered by a nurse, including symptom assessment and management, patient education on lung cancer and treatment options, discussion and communication about preferences for care, psychosocial assessment (including referrals to ancillary services), and patient-centered resources. A personalized treatment plan based on the patient's lung cancer stage, treatment, symptoms and psychosocial needs will be developed by the palliative care team (physician, study nurse) with input from the patient and family member. The study nurse will assess patient's symptoms, implement and monitor the treatment plan applying established End-of- Life Nursing Education Consortium (ELNEC) for Veterans protocols.
  Other Names: Supportive Care
  Arms: Intervention

SUMMARY:
The focus of the study is to test a nurse-led telephone-based palliative care intervention on improving the delivery of care for patients with newly diagnosed lung cancer. The study is a three site randomized control trial to determine the efficacy of the intervention on improving patients' quality of life, symptom burden, and satisfaction of care. Additionally, the study will test an innovative care delivery model to improve patients' access to palliative care. The investigators will also determine the effect of the intervention on patient activation to discuss treatment preferences with their clinician and on clinician knowledge of patients' goals of care.

DETAILED DESCRIPTION:
Patients meeting entry criteria will be randomized to the intervention arm, palliative care plus usual care, or the usual care arm. Patients randomized to the intervention arm will receive usual oncologic care and phone calls from a nurse. Outcome measures will be collected at baseline and at the end of the patients' primary cancer treatment. The study will be performed at the Puget Sound Health Care System, Birmingham VA and Portland VA. The investigators will recruit individuals (n=138) with lung cancer over 2.5 years. The primary objective is to determine the efficacy of the nurse-led telephone-based palliative intervention on improving patients' quality of life, symptom burden, and satisfaction of care. In addition, using validated instruments, the investigators will assess the effect of the intervention on patient activation to discuss treatment preferences with their clinician and on clinician knowledge of patients' goals of care. The results of this study will inform a future effectiveness/implementation study.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed at the Puget Sound Health Care System, Birmingham VA, or Portland VA with a primary diagnosis of lung cancer that requires more than surgical resection:

* diagnosed within 8 weeks of recruitment
* must have telephone access
* ability to understand English
* able to participate in informed consent process

Exclusion Criteria:

Patients not eligible to participate in the study include those who are inpatients prior to randomization,

* those who are under the care of palliative care or hospice at the time of randomization
* those who have severe mental health disorders
* those who are unable to speak directly with the nurse over the telephone
* or those that have the inability to provide informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn F. Reinke, PhD ARNP, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (3):
- United States (3):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reinke LF, Meier DE. Research Priorities in Subspecialty Palliative Care: Policy Initiatives. J Palliat Med. 2017 Aug;20(8):813-820. doi: 10.1089/jpm.2017.0303. PMID 28777716
- [Result] Aslakson RA, Reinke LF, Cox C, Kross EK, Benzo RP, Curtis JR. Developing a Research Agenda for Integrating Palliative Care into Critical Care and Pulmonary Practice To Improve Patient and Family Outcomes. J Palliat Med. 2017 Apr;20(4):329-343. doi: 10.1089/jpm.2016.0567. PMID 28379812
- [Result] Reinke LF, Vig EK, Tartaglione EV, Backhus LM, Gunnink E, Au DH. Protocol and pilot testing: The feasibility and acceptability of a nurse-led telephone-based palliative care intervention for patients newly diagnosed with lung cancer. Contemp Clin Trials. 2018 Jan;64:30-34. doi: 10.1016/j.cct.2017.11.013. Epub 2017 Nov 23. No abstract available. PMID 29175560
- [Result] Sullivan DR, Chan B, Lapidus JA, Ganzini L, Hansen L, Carney PA, Fromme EK, Marino M, Golden SE, Vranas KC, Slatore CG. Association of Early Palliative Care Use With Survival and Place of Death Among Patients With Advanced Lung Cancer Receiving Care in the Veterans Health Administration. JAMA Oncol. 2019 Dec 1;5(12):1702-1709. doi: 10.1001/jamaoncol.2019.3105. PMID 31536133
- [Result] Sullivan DR, Ganzini L, Delorit MA, Slatore CG, Vranas KC, Golden SE, Hansen L. Transcending silos and building relationships: A qualitative study of palliative care use and integration in a national health system. [Abstract]. American journal of respiratory and critical care medicine. 2020 Nov 1; 201(B22):A2820.
- [Result] Sullivan DR, Slatore CG, Stone K, Nugent S, Kern J, Farris M, Roszenweig K, Swanson S, J Wisnivesky JP. Associations between Treatment and Team Composition with Decisional Regret among Patients with Early Stage Lung Cancer. [Abstract]. American journal of respiratory and critical care medicine. 2020 Nov 1; 201(B22):A4726.
- [Result] Vranas KC, Plinke W, Bourne D, Kansagara D, Lee RY, Kross EK, Slatore CG, Sullivan DR. The influence of POLST on treatment intensity at the end of life: A systematic review. J Am Geriatr Soc. 2021 Dec;69(12):3661-3674. doi: 10.1111/jgs.17447. Epub 2021 Sep 22. PMID 34549418
- [Result] Hedstrom GH, Hooker ER, Howard M, Shull S, Golden SE, Deffebach ME, Gorman JD, Murphy K, Fabbrini A, Melzer AC, Slatore CG. The Chain of Adherence for Incidentally Detected Pulmonary Nodules after an Initial Radiologic Imaging Study: A Multisystem Observational Study. Ann Am Thorac Soc. 2022 Aug;19(8):1379-1389. doi: 10.1513/AnnalsATS.202111-1220OC. PMID 35167780

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We identified lung cancer patients at the Puget Sound Health Care System, the Birmingham VA, and the Portland VA. Virtually all patients undergoing evaluation for lung cancer were presented at the Tumor Board and/or were evaluated in the chest (thoracic surgery and pulmonary), oncology, radiation oncology, or lung cancer clinics. All patients were screened weekly to determine study eligibility. Recruitment began when the first patient enrolled on December 2016 and lasted to June 2019.
Pre-assignment Details: If consented participants became ineligible, they were not randomized into one of the two study arms.
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 73 | 78
Completed | 57 | 65
Not Completed | 16 | 13
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Death | 5 | 7
Not completed — Lost to Follow-up | 3 | 2
Not completed — Enrolled in Hospice | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 73 | 78 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean, SD
  years
    Age | 69.0 (8.6) | 70.0 (6.4) | 69.5 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 71 | 77 | 148
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 9 | 14
  White | 65 | 63 | 128
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Lung Total Outcome Index Score at Final Visit
Description: Patient Quality of Life including symptoms as measured by the FACT-L (Functional Assessment of Cancer Therapy-Lung Scale). The FACT-L outcome measure reported is the mean change in the TOI subscale (Total Outcome Index) of the instrument, computed as the differences between final and baseline visit scores. The TOI subscale range is 0-84, with a higher score indicating a better quality of life. Among patients with newly diagnosed lung cancer, provision of a telephone-based palliative care intervention will be associated with a change in FACT-L TOI score. The investigators will assess the difference in FACT-L TOI scores between the intervention and control subjects.
Time Frame: Baseline and 3 Months
Population: Difference in FACT-L TOI score, Final Visit Measure, minus Baseline Visit Measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 73 | 78
score on a scale | 1.8 (16.8) | -1.2 (13.2)

2. Secondary Outcome: Change From Baseline in Patient Satisfaction of Care at Final Visit
Description: Patient satisfaction with care will be assessed by using the FAMCARE-Patient Survey 13 (full unabbreviated scale name). The FAMCARE is a 13 item, 5 point likert-scale validated questionnaire measuring patient satisfaction with cancer care and assessing interactions with health care providers, performance status and symptom burden. Only total score are reported (no subscales). Scores range from 13-65 with scores of 52 > being satisfied with care. In full randomized clinical trials the estimated MID is 5 points from baseline to 12 weeks. Among patients with newly diagnosed lung cancer, provision of a telephone-based palliative care intervention will be associated with a change in FAMCARE-P13 score. The investigators will assess the difference in FAMCARE-P13 scores between the intervention and control subjects.
Time Frame: Baseline and 3 Months
Population: Difference in FAMCARE-13 Score, Final Visit measure minus Baseline Visit Measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 73 | 78
score on a scale | 1.1 (7.6) | 0.5 (8.2)

ADVERSE EVENTS:
Time Frame: Each participant was assessed for adverse events through the study completion, e.g. 3 months or at the end of cancer treatment.
Description: ER visits, hospitalizations, and death are expected for patients with advanced cancers. All ER/Hospitalizations/Deaths were collected during medical record review and patients self-report (intervention arm only). They were reviewed at weekly study meetings and annually by the IRBs for each study site. Organ systems were not collected. N/A
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 5/73 | 7/78
Serious Adverse Events (participants affected / at risk) | 19/73 | 11/78
Other Adverse Events (participants affected / at risk) | 22/73 | 13/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=73) | Usual Care (N=78)
Serious adverse events (Respiratory, thoracic and mediastinal disorders) | 19 (29) | 11 (14) — Hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=73) | Usual Care (N=78)
Emergency Department Visits (General disorders) | 22 (35) | 13 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT03007953/Prot_SAP_000.pdf